CLINICAL TRIAL: NCT01778036
Title: Neck Motion and Motor Control in Chronic Neck Pain and Associations With Clinical Symptoms
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Sponsor
Other Study IDs: 2011/2522
Record Dates: First submitted 2013-01-25; First posted 2013-01-29 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Neck Pain
Keywords: Neck movement; motor control; disability; psychological variables; Head Movements; Physical therapy; Fear avoidance; Self Efficacy; Catastrophizing; Fly test; Postural sway
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neck pain patients following physiotherapy treatment: Neck pain patients will follow physiotherapy treatment in primary health care.

SUMMARY:
The primary purpose of this study is to investigate if there is altered motor control of head and neck in chronic neck pain patients compared with healthy persons. In addition, associations between neck pain, motor control, disability and function, and clinical symptoms will be studied in patients following physiotherapy treatment in primary health care.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic neck pain with duration >2 weeks
* Normal or corrected vision
* Pain at or above 3 on Numeric Rating Scale, with "low pain" defined as 3-4 and "high pain" as 5 or higher.

Exclusion Criteria:

* Systemic or diagnosed chronic disease, including diabetes, stroke and neurological diseases, that may influence motor control and neck pain or ability to perform tests
* positive spurling test for neurological radiating arm pain
* pregnancy
* whiplash
* insufficient comprehension of Norwegian language

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neck pain patients referred to physiotherapy treatment in primary health care
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Conjunct motion | up to 8 weeks
  Describes the movement stiffness in active movements of the neck. Conjunct motion is movement in the two associated movement planes to the primary plane. For example,the amount of rotation and lateral flexion during neck flexion and extension. Measured by 3D Liberty device and with degrees as unit of measure.

SECONDARY OUTCOMES:
head motion smoothness | up to 8 weeks
  Measured by a 3D Liberty device and with velocity(degrees/s)as unit of measure
reposition accuracy | up to 8 weeks
  Measured by 3D Liberty device and with degrees as unit of measure
postural sway. | up to 8 weeks
  Measured by 3D Liberty device and trunk sway as a unit of measure
Head stabilization | up to 8 weeks
  Measured by 3D Liberty device and with velocity (degrees/second) as unit of measure
pain | up to 24 weeks
  a numerical pain rating scale will be used to measure neck pain.
Head motion accuracy | up to 8 weeks
  Head motion accuracy will be measured by a 3D Liberty device and centimeter will be used as a unit of measure

OTHER OUTCOMES:
Neck disability and function | up to 24 weeks
  Neck Disability Index and patient specific functional scale(Tampa Scale of Kinesiophobia, Pain Catastrophizing Scale and Pain Self Efficacy Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Ottar Vasseljen, prof, Study Director — Norwegian University of Science and Technology
Locations (2):
- Norway (2):
  - University of Oslo, Oslo
  - Norwegian University of Science and Technology, Trondheim

REFERENCES:
- [Result] Meisingset I, Stensdotter AK, Woodhouse A, Vasseljen O. Neck motion, motor control, pain and disability: A longitudinal study of associations in neck pain patients in physiotherapy treatment. Man Ther. 2016 Apr;22:94-100. doi: 10.1016/j.math.2015.10.013. Epub 2015 Nov 2. PMID 26586133